CLINICAL TRIAL: NCT02563626
Title: Coronary Artery Aneurysms: Incidence, Management and Long Term Prognosis
Brief Title: Coronary Artery Aneurysm Registry
Acronym: CAAR
Status: Completed | Type: Observational
Sponsor: St Carlos Hospital, Madrid, Spain (Other)
Responsible Party: Principal Investigator, IVAN J NUÑEZ GIL, MD, PhD, FESC, St Carlos Hospital, Madrid, Spain
Other Study IDs: CAAR
Record Dates: First submitted 2015-09-26; First posted 2015-09-30 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Aneurysm
Keywords: coronary artery aneurysm; prognosis; outcomes; management; incidence; heart failure; acute coronary syndrome; death
MeSH Terms: conditions — Coronary Aneurysm; Heart Failure; Acute Coronary Syndrome; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
International registry gathering patients with angiographically confirmed coronary aneurysm.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE:

Coronary artery aneurysm is defined as coronary dilatation which exceeds the diameter of normal adjacent segments or the diameter of the patient's largest coronary vessel by 1.5 times. Described by Bourgon, it is an uncommon disease which has been diagnosed with increasing frequency since the advent of coronary angiography. The incidence varies from 1.5% to 5% with male dominance and a predilection for the right coronary artery.

Although several causes have been reported, atherosclerosis accounts for 50% of coronary aneurysms in adults. Reported complications include thrombosis and distal embolization, rupture and vasospasm, causing ischemia, heart failure or arrhythmias. The natural history and prognosis remains obscure, since definitive data are scarce. Controversies persist regarding the use of medical management (antithrombotic) or interventional/surgical procedures.

OBJECTIVES.

Taking into account the classical coronary aneurysm definition, the investigators propose:

* ANATOMIC OBJECTIVES.

  * To characterize coronary aneurysms frequency over all cause invasive coronary angiography.
  * To describe anatomy, location and aneurysms features.
  * To assess intracoronary imaging data if available.
  * To describe the natural history, when evolutive chats were available
* CLINICAL OBJECTIVES.

  * Cause for the diagnostic catheterization and aneurysms symptoms, if present.
  * Patient´s clinical features.
  * Long-term outcomes.
* THERAPEUTIC OBJECTIVES.

  * To assess management strategies, conservative, interventional or surgical and its short and long term results.
  * Outcomes regarding management.

DESIGN:

* Retrospective recruitment, prospective follow-up registry.
* Multicentric/international.
* Anonymized.
* Electronic database. Centralized analysis (core) at Hospital Clínico San Carlos.
* Recruitment: 1/january/2002-1/december/2015.

ELIGIBILITY:
Inclusion Criteria (angiographic diagnosis):

* Coronary aneurysm: focal coronary dilatation which exceeds the diameter of normal adjacent segments or the diameter of the patient's largest coronary vessel by 1.5 times.

Exclusion Criteria:

* Patient ´s refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a coronary aneurysm diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1565 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Any cause death | 12 months
  dicotomic variable (yes/no)
Cardiology readmission | 12 months
  dicotomic variable (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: IVAN J NUÑEZ GIL, MD,PhD,FESC, Study Chair — HOSPITAL CLINICO SAN CARLOS.
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Background] SCOTT DH. Aneurysm of the coronary arteries. Am Heart J. 1948 Sep;36(3):403-21. doi: 10.1016/0002-8703(48)90337-8. No abstract available. PMID 18880707
- [Background] Swaye PS, Fisher LD, Litwin P, Vignola PA, Judkins MP, Kemp HG, Mudd JG, Gosselin AJ. Aneurysmal coronary artery disease. Circulation. 1983 Jan;67(1):134-8. doi: 10.1161/01.cir.67.1.134. PMID 6847792
- [Background] Syed M, Lesch M. Coronary artery aneurysm: a review. Prog Cardiovasc Dis. 1997 Jul-Aug;40(1):77-84. doi: 10.1016/s0033-0620(97)80024-2. PMID 9247557
- [Background] Dutary J, Zakhem B, DE Lucas CB, Paulo M, Gonzalo N, Alfonso F. Treatment of a giant coronary artery aneurysm: intravascular ultrasound and optical coherence tomography findings. J Interv Cardiol. 2012 Feb;25(1):82-5. doi: 10.1111/j.1540-8183.2011.00659.x. Epub 2011 May 22. PMID 21599751
- [Background] Maehara A, Mintz GS, Ahmed JM, Fuchs S, Castagna MT, Pichard AD, Satler LF, Waksman R, Suddath WO, Kent KM, Weissman NJ. An intravascular ultrasound classification of angiographic coronary artery aneurysms. Am J Cardiol. 2001 Aug 15;88(4):365-70. doi: 10.1016/s0002-9149(01)01680-0. PMID 11545755
- [Result] Nunez-Gil IJ, Nombela-Franco L, Bagur R, Bollati M, Cerrato E, Alfonso E, Liebetrau C, De la Torre Hernandez JM, Camacho B, Mila R, Amat-Santos IJ, Alfonso F, Rodriguez-Olivares R, Camacho Freire SJ, Lozano I, Jimenez Diaz VA, Piraino D, Latini RA, Feltes G, Linares JA, Mancone M, Ielasi A, Sanchez-Grande Flecha A, Fernandez Cisnal A, Ugo F, Jimenez Mazuecos JM, Omede P, Pavani M, Villablanca PA, Louka BF, Fernandez-Ortiz A; CAAR Investigators. Rationale and design of a multicenter, international and collaborative Coronary Artery Aneurysm Registry (CAAR). Clin Cardiol. 2017 Aug;40(8):580-585. doi: 10.1002/clc.22705. Epub 2017 Mar 24. PMID 28337781
- [Result] Nunez-Gil IJ, Cerrato E, Bollati M, Nombela-Franco L, Terol B, Alfonso-Rodriguez E, Camacho Freire SJ, Villablanca PA, Amat Santos IJ, de la Torre Hernandez JM, Pascual I, Liebetrau C, Camacho B, Pavani M, Albistur J, Latini RA, Varbella F, Jimenez-Diaz VA, Piraino D, Mancone M, Alfonso F, Linares JA, Rodriguez-Olivares R, Jimenez Mazuecos JM, Palazuelos Molinero J, Sanchez-Grande Flecha A, Gomez-Hospital JA, Ielasi A, Lozano I, Omede P, Bagur R, Ugo F, Medda M, Louka BF, Kala P, Escaned J, Bautista D, Feltes G, Salinas P, Alkhouli M, Macaya C, Fernandez-Ortiz A; CAAR investigators. Coronary artery aneurysms, insights from the international coronary artery aneurysm registry (CAAR). Int J Cardiol. 2020 Jan 15;299:49-55. doi: 10.1016/j.ijcard.2019.05.067. Epub 2019 Jul 19. PMID 31378382
- [Result] D'Ascenzo F, Saglietto A, Ramakrishna H, Andreis A, Jimenez-Mazuecos JM, Nombela-Franco L, Cerrato E, Liebetrau C, Alfonso-Rodriguez E, Bagur R, Alkhouli M, De Ferrari GM, Nunez-Gil IJ; CAAR Investigators. Usefulness of oral anticoagulation in patients with coronary aneurysms: Insights from the CAAR registry. Catheter Cardiovasc Interv. 2021 Nov 1;98(5):864-871. doi: 10.1002/ccd.29243. Epub 2020 Sep 9. PMID 32902099
- [Result] Arslan F, Nunez-Gil IJ, Rodriguez-Olivares R, Cerrato E, Bollati M, Nombela-Franco L, Terol B, Alfonso-Rodriguez E, Camacho Freire SJ, Villablanca PA, Amat Santos IJ, De la Torre Hernandez JM, Pascual I, Liebetrau C, Alkhouli M, Fernandez-Ortiz A; Coronary Artery Aneurysm Registry (CAAR) investigators. Sex differences in treatment strategy for coronary artery aneurysms: Insights from the international Coronary Artery Aneurysm Registry. Neth Heart J. 2022 Jun;30(6):328-334. doi: 10.1007/s12471-021-01649-5. Epub 2021 Dec 15. PMID 34910278